CLINICAL TRIAL: NCT01815762
Title: Extravascular Lung Water Monitoring by Combined Ultrasound and Bioimpedance as a Guide for Treatment in Hemodialysis Patients
Acronym: BUST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, MD, PhD, FRCP, Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RandBCM
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-03

CONDITIONS: Patients on Hemodialysis for More Than 3 Months
Keywords: bioimpedance; overhydration; hemodialysis; arterial stiffness; mortality
MeSH Terms: conditions — Water Intoxication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- active arm of the study (Active Comparator): The number of ultrasound lung comets (ULC) will directly adjust the prescribed post-hemodialysis dry weight. The US B-line score (BLS) will be measured before dialysis. In patients presenting moderate to severe lung congestion (≥15 BLS pre-dialysis) LUS measurements will be repeated once a week until the treatment goal was achieved (<15 BLS pre-dialysis) and once a month thereafter. monthly monitoring frequency will be adopted also in patients without pulmonary congestion (BLS <15). Patients without evidence of lung congestion at baseline who developed pulmonary congestion (≥ 15 BLS) during the trial will received the same treatment contemplated for those with lung congestion at baseline during the trial.
  Interventions: Other: Active arm
- Standard care arm (No Intervention): In the control arm of the study, the dry weight will be assessed only clinically.Patients in the control arm of the study will be followed up and managed strictly with standard criteria according to current recommendations (implying optimization of fluids volume control on the basis of clinical criteria and the use of carvedilol, ACE inhibitors/sartans whenever deemed necessary); the use of lung US / bioimpedance assistance was not allowed in these patients.

INTERVENTIONS:
Other: Active arm — In the active arm of the study, the number of ultrasound lung comets (ULC) will directly adjust the prescribed post-hemodialysis dry weight. See study flowchart on page 1.
  If the patient does not tolerate the intervention (as described above), he will continue the study in the "medication arm", where the actual intervention in stopped, and extra cardio-protective drugs are added to the medication.
  Arms: active arm of the study

SUMMARY:
Patients will be selected from the Dialisys Centers in Iasi, Romania. Patients will be randomized 1:1 to have a dry-weight assessment based on clinical (control) or lung US and bioimpedance (active) guided protocol. In the control group post-dialysis dry weight will be adjusted based on clinical criteria only (blood pressure, presence of edema, intradialytic hypotension, cramps etc.) and in the active group the target weight will be prescribed using lung US and bioimpedance evaluation.

In patients randomized to the active arm of the study, the US B-line score (BLS) will be measured before dialysis and these measurements will be used to titrate ultrafiltration prescription. In patients presenting moderate to severe lung congestion (≥15 BLS pre-dialysis) LUS measurements will be repeated once a week until the treatment goal was achieved (<15 BLS pre-dialysis) and once a month thereafter. The same (monthly) monitoring frequency will be adopted also in patients without pulmonary congestion at pre-dialysis baseline (<15 BLS). Furthermore, the use of the technique is allowed whenever its application is deemed useful to assume clinical decisions by attending physicians. Patients in the active arm of the study without evidence of lung congestion at baseline who developed pulmonary congestion (≥ 15 BLS) during the trial will received the same treatment contemplated for those with lung congestion at baseline during the trial. The treatment goal will be pursued by ultrafiltration intensification realized within the same HD schedule (3 sessions x 4 hours/week) or, if not tolerated, by extra-dialyses, according to individual tolerance and feasibility. In case of clinical hypovolemia (persistent cramps, hypotension etc) additional dry-weight adjustments will be performed according to the bioimpedance measurement, provided that the patients are below 15 BLS. This addition will be necessary in order to be able to increase the dry-weight in patients with a persistent BLS < 15 and avoid under perfusion.

Patients in the control arm of the study will be followed up and managed strictly with standard criteria according to current recommendations (implying optimization of fluids volume control on the basis of clinical criteria and the use of carvedilol, ACE inhibitors/sartans whenever deemed necessary); the use of lung US / bioimpedanc assistance will not be messured in these patients.

The main exclusion criteria will be the presence of severe cardiac failure (NYHA class III-IV), past myocardial infarction, stable or unstable angina and acute coronary syndrome. Due to bioimpedance assessment limitation patients with metallic joint prostheses, cardiac stent or pacemakers, decompensated cirrhosis, pregnancy and limb amputations will be excluded, as BIS cannot be accurately performed in such cases. Due to lung US measurement limitation we will exclude patients with known persistent pleurisy, pulmonary fibrosis or pneumectomy. Other exclusion criteria will be malignancy, active infections, temporary or permanent catheter as a vascular access, mental incompetence and unwillingness to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* patients in hemodialysis for more than 3 months, that have no absolute contraindication for for performing bioimpedance measurements (amputation, stent, pregnancy, severe ascites) and ultrasound lung comets measurements (persistent pleuresia, pulmonary fibrosis, pneumectomy).

Exclusion Criteria:

* Patients with metallic joint prostheses, cardiac pacemakers, decompensated cirrhosis, limb amputations and severe conditions with life expectations <1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2013-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 2 years

SECONDARY OUTCOMES:
Left ventricular mass measured by echocardiography | 2 years

OTHER OUTCOMES:
Volume measures | 2 years
  bio-impedance (RXc graph, vector length, impedance ratio, phase angle, ECW:TBW ratio), weight, N-BNP, mean and pulse arterial pressure
Health-related quality of life (HRQOL) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Covic, MD, PhD, FRCP, Principal Investigator — University of Medicine and Pharmacy "Gr. T. Popa", Iasi, Nephrology Department
Locations (1):
- University Hospital "Dr. C.I. Parhon", Iasi, Department of Nephrology, Iași, Iaşi, Romania